CLINICAL TRIAL: NCT02491606
Title: Evaluation of Weekly Tafenoquine (SB 252263 / WR 238605) Compared to Placebo for Chemosuppression of Plasmodium Falciparum in Western Kenya
Brief Title: Evaluation of Weekly Tafenoquine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: SmithKline Beecham (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-7540
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — tafenoquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Load only (Experimental): Loading with tafenoquine 400 mg base for three days followed by placebo weekly.
  Interventions: Drug: Tafenoquine
- Low weekly dose (Experimental): Loading with tafenoquine 200 mg base for 3 days followed by tafenoquine 200 mg weekly.
  Interventions: Drug: Tafenoquine
- High weekly dose (Experimental): Loading with tafenoquine to 400 mg base for 3 days followed by tafenoquine 400 mg base weekly.
  Interventions: Drug: Tafenoquine
- Placebo (Experimental): Loading with placebo for 3 days followed by placebo once weekly.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine 200mg and 400 mg
  Arms: High weekly dose; Load only; Low weekly dose
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a phase 2b, placebo controlled, randomized, blinded study of the efficacy of WR 238605, a new primaquine analog, compared to placebo as chemosuppression of P. falciparum malaria in Nyanza Province, western Kenya.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects (male or female)
2. Age of 18-55 years
3. Residing in one of the study villages of the Nyanza Province for the entire study

Exclusion Criteria:

1. Any cardiovascular, liver, neurologic, or renal functional abnormality which in the opinion of the clinical investigators would place the subject at increased risk of an adverse event or confuse the result.
2. Female subjects who were pregnant (Positive serum / plasma -HCG as tested within 48 hours of first drug administration).
3. Use of antimalarial drugs not prescribed by study physicians within 2 weeks of study drug initiation.
4. Clinically significant abnormalities (including but not limited to abnormal hepatic or renal function) as determined by history, physical and routine blood chemistries and complete blood count.
5. Known hypersensitivity to any study drug.
6. Unwilling to remain in area and report for drug administration and blood drawing during the duration of the study.
7. Glucose 6 Phosphate Dehydrogenase (G6PD) deficiency.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 249 (Actual)
Dates: Start 1997-05; Primary Completion 1997-09 (Actual); Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Prophylactic outcome. | 13 Weeks
  Thick blood films were stained with Giemsa stain and malaria parasite counts determined by counting the number of asexual parasites per 200 white blood cells.
  A blood slide was not considered negative until an examination of 200 oil immersion fields showed no parasites.

SECONDARY OUTCOMES:
Prophylactic outcome after 7 weeks | 7 Weeks
  Thick blood films were stained with Giemsa stain and malaria parasite counts determined by counting the number of asexual parasites per 200 white blood cells.
  A blood slide was not considered negative until an examination of 200 oil immersion fields showed no parasites.
Prophylactic outcome after 10 weeks | 10 Weeks
  Thick blood films were stained with Giemsa stain and malaria parasite counts determined by counting the number of asexual parasites per 200 white blood cells.
  A blood slide was not considered negative until an examination of 200 oil immersion fields showed no parasites.

CONTACTS AND LOCATIONS:
Overall Officials: A.J Oloo, Principal Investigator — Kenya Medical Research Institute

REFERENCES:
- [Derived] Novitt-Moreno A, Ransom J, Dow G, Smith B, Read LT, Toovey S. Tafenoquine for malaria prophylaxis in adults: An integrated safety analysis. Travel Med Infect Dis. 2017 May-Jun;17:19-27. doi: 10.1016/j.tmaid.2017.05.008. Epub 2017 May 8. PMID 28495354